CLINICAL TRIAL: NCT00822965
Title: Patient Knowledge of Pacemaker/Implantable Cardioverter-Defibrillator-Phase II
Brief Title: Enhancing Knowledge Implantable Cardioverter-Defibrillators (ICDs)
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Mike Hogg Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2008-0163
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Pacemaker; Implantable Cardioverter-Defibrillators
Keywords: Pacemakers; PM; Implantable cardioverter-defibrillators; ICD; Implantable pulse generators; Educational Interventions
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient Knowledge Assessments: Questionnaires + Phone Interview
  Interventions: Other: Questionnaires; Other: Phone Interviews; Behavioral: Educational Packet

INTERVENTIONS:
Other: Questionnaires — 3 sets of questionnaires at the beginning of the study, at 2-months and at 4-months.
  Other Names: Survey
Other: Phone Interviews — 2 follow-up phone interviews.
Behavioral: Educational Packet — Video or DVD of device information, updates, recalls, on-line resources and benefits of routine follow-up for device(s).

SUMMARY:
The specific aims of the patient intervention are to:

1. increase patient knowledge about pacemakers (PM) and implantable cardioverter-defibrillators (ICDs)
2. help patients to identify if their PM or ICD has been interrogated
3. improve patient's physician-patient communication skills
4. teach patients how to identify if their device has been recalled
5. train patients what to do in case of a device recall

The educational interventions proposed, if proven to be effective by this pilot, will provide a low-cost, reproducible intervention to improve the clinical care and safe management of pacemakers (PM) and implantable cardioverter-defibrillators (ICD) in patients. The goal of the intervention will be to promote the safe use of implantable pulse generators.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will complete 3 sets of questionnaires (at the beginning of the study, at 2-months and at 4-months) which will be sent to you and returned by you through the mail. This will not require you to travel to M.D. Anderson. In addition to the questionnaires, you will also complete 2 follow-up phone interviews.

Questionnaires:

The first set of questionnaires will be mailed to your home. The questionnaires will ask questions about your anxiety level and how much you know about pacemakers or implantable cardioverter-defibrillators. There will also be questions about your gender, age, ethnicity, and race. The questionnaires will take about 25 minutes to complete. When you are finished, you will mail the questionnaires to the study staff. An envelope with pre-paid postage will be provided.

Educational Packet:

After you have completed the questionnaires, you will receive an educational packet in the mail. The packet will have a DVD or a video (depending on whether you tell us you have a DVD player or a VHS player) with information on medical devices, device recall information (when and why certain devices have been recalled in the past), a list of on-line resources and benefits of routine follow-up.

Phone Interview:

The study staff will call your home 1 week after you receive the educational packet for a follow-up interview. A member of the study staff will review the packet with you. The phone call will last about 20 minutes.

Additional Questionnaires:

Approximately 2 months and at 4 months after you complete the first set of questionnaires, an additional set of questionnaires will be mailed to you. You will be asked to complete the same questionnaires as you did in the first set. At 4 months an additional questionnaire about the information in the educational packet and how useful it was to you will be included. The questionnaires will take about 25 minutes to complete. When you are finished, you will mail the questionnaires to the study staff. An envelope with pre-paid postage will be provided.

Length of Study:

You participation on this study is complete once you have completed the additional questionnaires.

This is an investigational study. Up to 104 patients will be enrolled in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients (beginning with most recent date) who presented to UTMDACC Preoperative Consultation Clinic from January 1, 2000 to November 15, 2008 with an implanted pulse generator.
2. English-speaking (Resources to translate materials and provide interviews in Spanish language or languages other than English are not available for this study).
3. Adult patients 18 years of age or older.

Exclusion Criteria:

1. Patients who fail to consent to participate.
2. Patients with self-report of hearing impairment, sight, or reading impairment that would hinder ability to complete written surveys
3. Patients who have a second implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presented to UTMDACC Preoperative Consultation Clinic from January 1, 2000 to November 15, 2008 with an implanted pulse generator.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2009-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Patient knowledge about pacemakers (PM) and implantable cardioverter-defibrillators (ICDs) | Total knowledge score evaluated at baseline and at 2-month and 4-month post educational intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Suarez-Almazor, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org